CLINICAL TRIAL: NCT03155893
Title: A Randomized, Double-blind, Double-dummy, Placebo- and Positive-controlled Study to Evaluate the Cardiac Safety of a Single Dose of AL-335 Administered on a Background of Simeprevir and Odalasvir and of Repeated Doses of Odalasvir Administered Alone in Healthy Subjects
Brief Title: A Study to Evaluate the Cardiac Safety of a Single Dose of AL-335 Administered on a Background of Simeprevir and Odalasvir and of Repeated Doses of Odalasvir Administered Alone in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108332; 64294178HPC1012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Desvenlafaxine Succinate; adafosbuvir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Panel 1: Treatment A (Experimental): Participants will receive odalasvir (ODV) placebo (matching 25 milligram [mg] ODV [1*25 mg tablet]) and simeprevir (SMV) placebo (matching 150 mg SMV [2*75 mg capsules]) once daily from Day 1 to 16 along with single dose of AL-335 placebo (matching 1200 milligram [mg] AL-335 [3*400 mg tablets]) on Day 15 and moxifloxacin placebo (matching 400 mg moxifloxacin [1*400 mg capsule]) as a single dose on Day 1, 15 and 16 along with moxifloxacin 400 mg (1*400 mg capsule) single dose on Day 2 orally under fed conditions.
  Interventions: Drug: ODV Placebo (Matching 25 mg ODV); Drug: SMV Placebo (Matching 150 mg SMV); Drug: AL-335 Placebo (matching 1200 mg AL-335); Drug: Moxifloxacin Placebo (matching 400 mg moxifloxacin)
- Panel 1: Treatment B (Experimental): Participants will receive odalasvir (ODV) placebo (matching 25 milligram [mg] ODV [1*25 mg tablet]) and simeprevir (SMV) placebo (matching 150 mg SMV [2*75 mg capsules]) once daily from Day 1 to 16 along with single dose of AL-335 placebo (matching 1200 milligram [mg] AL-335 [3*400 mg tablets]) on Day 15 and moxifloxacin placebo (matching 400 mg moxifloxacin [1*400 mg capsule]) as a single dose on Day 1, 2 and 15 along with moxifloxacin 400 mg (1*400 mg capsule) single dose on Day 16 orally under fed conditions.
  Interventions: Drug: ODV Placebo (Matching 25 mg ODV); Drug: SMV Placebo (Matching 150 mg SMV); Drug: AL-335 Placebo (matching 1200 mg AL-335); Drug: Moxifloxacin Placebo (matching 400 mg moxifloxacin)
- Panel 1: Treatment C (Experimental): Participants will receive odalasvir (ODV) placebo (matching 25 milligram [mg] ODV [1*25 mg tablet]) and simeprevir (SMV) placebo (matching 150 mg SMV [2*75 mg capsules]) once daily on Day 1 and moxifloxacin placebo (matching 400 mg moxifloxacin [1*400 mg capsule]) as a single dose on Day 1, 2, 15 and 16 along with ODV 25 mg (1*25 mg tablet) and SMV 150 mg (2*75 mg capsule) once daily on Day 2 to 16 and AL-335 1200 mg (3*400 mg tablet) single dose on Day 15 orally under fed conditions.
  Interventions: Drug: ODV Placebo (Matching 25 mg ODV); Drug: SMV Placebo (Matching 150 mg SMV); Drug: Moxifloxacin Placebo (matching 400 mg moxifloxacin); Drug: ODV 25 mg; Drug: SMV 150 mg; Drug: AL-335 1200 mg
- Panel 2: Treatment E (Placebo Comparator): Participants will receive ODV placebo (matching 200 mg ODV [4*50 mg tablets]) on Days 1 and 2; ODV placebo (matching 125 mg ODV [2*50 mg tablets + 1*25 mg tablets]) on Days 3 to 7; and ODV placebo (matching 100 mg ODV [2*50 mg tablets] on Days 8 to 14, orally once daily under fed conditions.
  Interventions: Drug: ODV Placebo (Matching 200 mg ODV); Drug: ODV Placebo (Matching 125 mg ODV); Drug: ODV Placebo (Matching 100 mg ODV)
- Panel 2: Treatment F (Experimental): Participants will receive ODV 200 mg (4*50 mg tablets) on Days 1 and 2; ODV 125 mg (2*50 mg tablets + 1*25 mg tablets) on Days 3 to 7, and ODV 100 mg (2*50 mg tablets) on Days 8 to 14, orally once daily under fed conditions.
  Interventions: Drug: ODV 200 mg; Drug: ODV 125 mg; Drug: ODV 100 mg

INTERVENTIONS:
Drug: ODV Placebo (Matching 25 mg ODV) — Participants will receive ODV placebo (matching 25 [mg] ODV [1*25 mg tablet]) once daily in Treatment A and B from Day 1 to 16 and Treatment C on Day 1.
  Arms: Panel 1: Treatment A; Panel 1: Treatment B; Panel 1: Treatment C
Drug: ODV Placebo (Matching 200 mg ODV) — Participants will receive ODV placebo (matching 200 mg ODV [4*50 mg tablets]) on Days 1 and 2 in Treatment E.
  Arms: Panel 2: Treatment E
Drug: ODV Placebo (Matching 125 mg ODV) — Participants will receive ODV placebo (matching 125 mg ODV [2*50 mg tablets + 1*25 mg tablets]) orally once daily on Days 3 to 7 in Treatment E.
  Arms: Panel 2: Treatment E
Drug: ODV Placebo (Matching 100 mg ODV) — Participants will receive ODV placebo (matching 100 mg ODV [2*50 mg tablets] orally once daily on Days 8 to 14 in Treatment E.
  Arms: Panel 2: Treatment E
Drug: SMV Placebo (Matching 150 mg SMV) — Participants will receive SMV Placebo (matching 150 mg SMV [2*75 mg capsules]) orally once daily administered from Day 1 to 16 in Treatment A, B and on Day 1 in Treatment C.
  Arms: Panel 1: Treatment A; Panel 1: Treatment B; Panel 1: Treatment C
Drug: AL-335 Placebo (matching 1200 mg AL-335) — Participants will receive a single dose of AL-335 placebo (matching 1200 mg AL-335 [3*400 mg tablets]) administered orally on Day 15 in Treatment A and B.
  Arms: Panel 1: Treatment A; Panel 1: Treatment B
Drug: Moxifloxacin Placebo (matching 400 mg moxifloxacin) — Participants will receive a single dose of moxifloxacin placebo (matching 400 mg moxifloxacin [1*400 mg capsule]) administered orally on Day 1, 15 and 16 in Treatment A, on Day 1, 2 and 15 in Treatment B and on Day 1, 2, 15 and 16 in Treatment C.
  Arms: Panel 1: Treatment A; Panel 1: Treatment B; Panel 1: Treatment C
Drug: ODV 25 mg — Participants will receive ODV 25 mg orally once daily administered on Days 2 to 16 in Treatment C.
  Arms: Panel 1: Treatment C
Drug: ODV 200 mg — Participants will receive ODV 200 mg (4*50 mg tablets) orally once daily will be administered on Days 1 and 2 in Treatment F.
  Arms: Panel 2: Treatment F
Drug: ODV 125 mg — Participants will receive ODV 125 mg (2*50 mg tablets + 1*25 mg tablets) once daily administered on Days 3 to 7 in Treatment F.
  Arms: Panel 2: Treatment F
Drug: ODV 100 mg — Participants will receive ODV 100 mg (2*50 mg tablets) orally once daily administered on Days 8 to 14 in Treatment F.
  Arms: Panel 2: Treatment F
Drug: SMV 150 mg — Participants will receive SMV 150 mg (2*75 mg capsules) orally once daily administered on Days 2 to 16 in Treatment C.
  Arms: Panel 1: Treatment C
Drug: AL-335 1200 mg — Participants will receive a single oral dose of AL-335 1200 mg (3*400 mg tablets) administered on Day 15 in Treatment C.
  Arms: Panel 1: Treatment C

SUMMARY:
The main purpose of this study is to assess the effect of a single supratherapeutic dose of AL-335 administered on top of multiple doses of odalasvir (ODV) and simeprevir (SMV) versus placebo on QT/QT interval corrected for heart rate (QTc) interval changes, using intersection-union test (IUT) analysis (Panel 1); to assess the effect of ODV on QT/QTc and PR interval changes after multiple supratherapeutic doses of ODV using an exposure-response (ER) approach (Panel 2); and to assess the effect of multiple supratherapeutic doses of ODV on echocardiographic left ventricular ejection fraction (LVEF) (Panel 2) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign and date an informed consent form (ICF) indicating that he or she understands the purpose of, and the procedures required for, the study and is willing to participate in the study
* Participant must be healthy on the basis of physical examination, medical history, vital signs, and laboratory tests performed at screening
* Participant must have a blood pressure (supine after at least 5 minutes rest) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Participant must have a 12-lead electrocardiogram (ECG) (based on the mean value of triplicate ECG parameters) consistent with normal cardiac conduction and function at screening
* Participant must have an echocardiogram at screening with left ventricular ejection fraction (LVEF) greater than or equal to (>=)55 percent (%). Participant should not have any other echocardiogram finding suggestive of clinically relevant cardiomyopathy
* Female participant must have a negative highly sensitive urine pregnancy test at Day -2 (Panel 1) or Day -4 (Panel 2)

Exclusion Criteria:

* Participant has a history of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, constipation, or gastrointestinal surgery that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participant with a history of clinically relevant heart rhythm disturbances including atrial, junctional, re-entry, and ventricular tachycardia, and heart blocks
* Participant with unusual T-wave morphology (such as bifid T-wave) likely to interfere with corrected QT (QTc) measurements
* Participant with a past history of sick sinus syndrome, heart arrhythmias (example, extrasystolic rhythms or tachycardia at rest). Isolated extrasystolic beats are not exclusionary; risk factors associated with Torsade de Pointes (TdP) such as hypokalemia; family history of short/long QT syndrome; sudden unexplained death (including sudden infant death syndrome in a first-degree relative [that is, sibling, offspring, or biological parent])
* Participant with any skin condition likely to interfere with electrocardiogram (ECG) electrode placement or adhesion
* Participant with a breast implant or a history of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Panel 1:Effect of AL-335 Single Supratherapeutic Dose on QT/QTc Interval Change on top of Multiple Doses of ODV and SMV Vs. Placebo Using IUT Analysis at Day 16 | Baseline (Day 1), Day 15
  Intersection-union test (IUT) analysis will be performed to evaluate the effect of AL-335 on QT/QTc interval changes after a single supratherapeutic dose of AL-335 on top of multiple doses of odalasvir (ODV) and simeprevir (SMV) versus placebo.
Panel 2: Effect of ODV on QT/QTc Interval Change From Baseline After Multiple Supratherapeutic Doses of ODV Using ER Approach at Day 14 | Baseline (Day -3), Day 14
  Exposure-response (ER) analysis will be performed to evaluate the effect of ODV on QT/QTc interval changes after multiple supratherapeutic doses of ODV.
Panel 2: Effect of ODV on QT/QTc Interval Change From Baseline After Multiple Supratherapeutic Doses of ODV Using ER Approach at Day 15 | Baseline (Day -3), Day 15
  ER analysis will be performed to evaluate the effect of ODV on QT/QTc interval changes after multiple supratherapeutic doses of ODV.
Panel 2: Effect of ODV on QT/QTc Interval Change From Baseline After Multiple Supratherapeutic Doses of ODV Using ER Approach at Day 16 | Baseline (Day -3), Day 16
  ER analysis will be performed to evaluate the effect of ODV on QT/QTc interval changes after multiple supratherapeutic doses of ODV.
Panel 2: Effect of ODV on PR Interval Change From Baseline After Multiple Supratherapeutic Doses of ODV Using ER Approach at Day 14 | Baseline (Day -3), Day 14
  ER analysis will be performed to evaluate the effect of ODV on PR interval changes after multiple supratherapeutic doses of ODV.
Panel 2: Effect of ODV on PR Interval Change From Baseline After Multiple Supratherapeutic Doses of ODV Using ER Approach at Day 15 | Baseline (Day -3), Day 15
  ER analysis will be performed to evaluate the effect of ODV on PR interval changes after multiple supratherapeutic doses of ODV.
Panel 2: Effect of ODV on PR Interval Change From Baseline After Multiple Supratherapeutic Doses of ODV Using ER Approach at Day 16 | Baseline (Day -3), Day 16
  ER analysis will be performed to evaluate the effect of ODV on PR interval changes after multiple supratherapeutic doses of ODV.
Panel 2: Effect of Multiple Supratherapeutic Doses of ODV on Change From Baseline in Echocardiographic Left Ventricular Ejection Fraction (LVEF) at Day 10 | Baseline (Day -2 and -1), Day 10
  Echocardiogram measurements will be performed to evaluate the effect of multiple supratherapeutic doses of ODV on change in echocardiographic LVEF. The baseline for echocardiographic LVEF will be the average of Days -2 and -1.
Panel 2: Effect of Multiple Supratherapeutic Doses of ODV on Change From Baseline in Echocardiographic Left Ventricular Ejection Fraction (LVEF) at Day 14 | Baseline (Day -2 and -1), Day 14
  Echocardiogram measurements will be performed to evaluate the effect of multiple supratherapeutic doses of ODV on change in echocardiographic LVEF. The baseline for echocardiographic LVEF will be the average of Days -2 and -1.
Panel 2: Effect of Multiple Supratherapeutic Doses of ODV on Change From Baseline in Echocardiographic Left Ventricular Ejection Fraction (LVEF) at Day 28 | Baseline (Day -2 and -1), Day 28
  Echocardiogram measurements will be performed to evaluate the effect of multiple supratherapeutic doses of ODV on change in echocardiographic LVEF. The baseline for echocardiographic LVEF will be the average of Days -2 and -1.

SECONDARY OUTCOMES:
Panel 1: Maximum Observed Analyte Concentration (Cmax) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  The Cmax is the maximum observed analyte concentration.
Panel 1: Time to Reach the Maximum Observed Analyte Concentration (Tmax) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Panel 1: Area Under the Analyte Concentration-time Curve From Time 0 to 24 Hours Postdose (AUC24) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  AUC24 is defined as area under the analyte concentration-time curve from time 0 to 24 hours postdose.
Panel 1: Area Under the Analyte Concentration-time Curve from Time 0 to the Time of the Last Measurable Concentration (AUClast) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  AUClast is defined as area under the analyte concentration-time curve from time 0 to the time of the last measurable (non-below quantification limit [BQL]) concentration.
Panel 1: Apparent Terminal Elimination Half-life (t1/2term) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  Apparent terminal elimination half-life is defined as 0.693/lambda(z).
Panel 1: Apparent Terminal Elimination Rate Constant (Lambda[z]) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  Lambda(z) is defined as apparent terminal elimination rate constant, determined by linear regression using the terminal log-linear phase of the log transformed concentration versus time curve.
Panel 1: Area Under the Analyte Concentration-time Curve From Time 0 to Infinite Time (AUC[0-infinity]) of AL-335 and its 2 metabolites ALS-022399 and ALS-022227 | Panel 1, Day 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  The AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Panel 1 and 2: Maximum Observed Analyte Concentration (Cmax) of ODV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose; Panel 2, Day 14: predose, 1, 3, 4, 5, 6, 7, 8, 10, 12, 24, 28, 32, 36, 48, 52, 56, 60, and 72 hours postdose
  The Cmax is the maximum observed analyte concentration.
Panel 1 and 2: Time to Reach the Maximum Observed Analyte Concentration (Tmax) of ODV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose; Panel 2, Day 14: predose, 1, 3, 4, 5, 6, 7, 8, 10, 12, 24, 28, 32, 36, 48, 52, 56, 60, and 72 hours postdose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Panel 1 and 2: Minimum Observed Analyte Concentration (Cmin) of ODV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose; Panel 2, Day 14: predose, 1, 3, 4, 5, 6, 7, 8, 10, 12, 24, 28, 32, 36, 48, 52, 56, 60, and 72 hours postdose
  The Cmin is a minimum observed analyte concentration.
Panel 1 and 2: Observed Analyte Concentration Just Prior to the Beginning of a Dosing Interval (Ctrough) of ODV | Panel 1: Predose on Days 14 and 15; Panel 2: Predose on Day 14
  The Ctrough is the observed analyte concentration just prior to the beginning of a dosing interval.
Panel 1 and 2: Area Under the Analyte Concentration-time Curve From Time 0 to 24 hours Postdose (AUC24) of ODV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose; Panel 2, Day 14: predose, 1, 3, 4, 5, 6, 7, 8, 10, 12 and 24 hours postdose
  AUC24 is defined as area under the analyte concentration-time curve from time 0 to 24 hours postdose.
Panel 2: Observed Analyte Concentration of ODV | Panel 2, Days 10 and 14: 6 and 8 hours postdose; Day 28: 6 and 8 hours
  Observed analyte concentration of ODV will be assessed on Days 10, 14 and 28.
Panel 1: Maximum Observed Analyte Concentration (Cmax) of SMV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  The Cmax is the maximum observed analyte concentration.
Panel 1: Time to Reach the Maximum Observed Analyte Concentration (Tmax) of SMV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  The tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Panel 1: Minimum Observed Analyte Concentration (Cmin) of SMV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  The Cmin is the minimum observed analyte concentration.
Panel 1: Observed Analyte Concentration Just Prior to the Beginning of a Dosing Interval (Ctrough) of SMV | Panel 1: Predose on Days 14 and 15
  The Ctrough is the observed analyte concentration just prior to the beginning of a dosing interval.
Panel 1: Area Under the Analyte Concentration-time Curve From Time 0 to 24 hours Postdose (AUC24) of SMV | Panel 1, Days 14 and 15: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 24 hours postdose
  AUC24 is defined as area under the analyte concentration-time curve from time 0 to 24 hours postdose.
Panel 1 and 2: Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 49 (Panel 1) and Day 66 (Panel 2)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Panel 1: Effect of Moxifloxacin on the QT/QTc Interval Change From Baseline at Day 2 and 16 | Baseline (Day 1), Days 2 and 16
  The effect of moxifloxacin on the QT/QTc Interval changes will be assessed for assay sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States